CLINICAL TRIAL: NCT06432543
Title: Polyethylene Wear Particle Analysis of Total Hip Arthroplasty -International Multicenter Study-
Brief Title: Polyethylene Wear Particle Analysis of THA
Status: Recruiting | Type: Observational
Sponsor: Osaka Metropolitan University (Other)
Collaborators: Mayo Clinic (Other); Hospital for Special Surgery, New York (Other); Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Yukihide Minoda, Associate Professor, Osaka Metropolitan University
Other Study IDs: OMU 2023-132
Record Dates: First submitted 2024-05-16; First posted 2024-05-29 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Wear of Articular Bearing Surface of Prosthetic Joint; Hip Arthropathy
Keywords: Polyethylene wear particle; Total hip arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The pericapsular tissue, which is removed during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- polyethylene containing Vitamin E: polyethylene containing Vitamin E
  Interventions: Device: polyethylene
- conventional polyethylene (no highly cross-linking): conventional polyethylene (no highly cross-linking)
  Interventions: Device: polyethylene
- conventional polyethylene (with highly cross-linking): conventional polyethylene (with highly cross-linking)
  Interventions: Device: polyethylene

INTERVENTIONS:
Device: polyethylene — No intervention as this is an observational study

SUMMARY:
Purpose of research The purpose of this study was to demonstrate that polyethylene (Vitamin E-containing polyethylene), a newly introduced biomaterial for tibial inserts in hip replacement surgery and widely used clinically, but whose mid- to long-term clinical results are still unknown, is superior to conventional polyethylene in vivo. The aim of this project is to conduct an international multi-center joint research study to determine whether polyethylene wear debris production can be reduced in the future, using an in vivo polyethylene wear debris analysis method that the investigators developed as a method that can provide early feedback.

DETAILED DESCRIPTION:
Research method In this study, the investigators conducted the following steps to determine the in vivo wear particles (number, size, and morphology) of conventional polyethylene, whose long-term results have already been clarified, and vitamin E-containing polyethylene, whose mid- to long-term results have not yet been clarified. Clarifying the difference.

Target of this research In this study, the investigators will focus on patients undergoing revision hip arthroplasty as a routine medical treatment.

First total joint replacement

* 30 patients using polyethylene containing Vitamin E
* 30 patients using conventional polyethylene (no high cross-linking)
* 30 patients using conventional polyethylene (with high cross-linking)

Accumulation of periarticular tissue In this study, the investigators will focus on patients undergoing revision hip arthroplasty as a routine medical treatment.

The test will be conducted after obtaining approval from the ethics committee at each facility and obtaining informed consent. The pericapsular tissue, which is removed during surgery and usually discarded, is obtained and fixed in formalin fixative. The tissue will be transported to the Department of Orthopedic Surgery, Osaka Public University Graduate School of Medicine for analysis. International transportation of tissues requires outsourcing to specialized companies with experience in transporting tissues from overseas.

Isolation of polyethylene wear debris The collected tissue around the joint capsule is immersed in 5Mol sodium hydroxide at 65°C for 1 hour to decompose the protein. Make a sucrose layer (5, 10, 20%) in a 14ml tube (14PA tube, Hitachi Koki Co, Ltd, Tokyo, Japan), add the dissolved solution, and place in an ultracentrifuge (CP100a, P28S1014 rotor, Hitachi Koki). Ultracentrifuge at 28,000 rpm [103,7009g] for 3 hours at 4°C. Prepare an isopropanol layer (0.90 and 0.96 g/mL) in a 40 ml tube (40PA tube, Hitachi Koki Co, Ltd, Tokyo, Japan), add the upper layer of sucrose layer, and centrifuge at 28,000 rpm (103,7009 g) and perform ultracentrifugation at 4°C for 1 hour. The isopropanol interlayer is collected to isolate polyethylene wear debris.

Analysis of polyethylene wear debris The isopropanol interlayer is filtered through a 0.1 μm polycarbonate filter (VCTP 013-00, Millipore Corporation, Bedford, MA). Dry the polycarbonate filter, fix it on an aluminum pedestal (M4, Nisshin EM Co, Ltd, Tokyo, Japan), and apply platinum coating (E-1030 ion sputter, Hitachi Science Systems Ltd, Tokyo, Japan). Observe the polyethylene wear particles on the polycarbonate filter using a scanning electron microscope (S4700SI, Hitachi Ltd, Tokyo, Japan), and analyze the following items using an image analyzer (Mac Scope, Mitani Co, Tokyo, Japan).

* Number of polyethylene wear particles (number per 1g of tissue)
* Size (Equivalent circle diameter [μm])
* Shape (aspect ratio, roundness)

Comparison of iv vivo polyethylene wear powder morphology depending on polyethylene material The number, size, and form of polyethylene wear debris will be compared between conventional polyethylene, whose long-term results have already been clarified, and vitamin E-containing polyethylene, whose medium- to long-term results have not yet been clarified. The investigators also investigated factors that affect polyethylene wear in vivo (age, height, weight, period from initial surgery to revision surgery, hip joint range of motion, hip prosthesis clinical score [Hip dysfunction and Osteoarthritis Outcome Score for Joint Replacement [HOOS Jr], Harris Hip Score, University of California Los Angeles [UCLA] activity score]).

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing revision hip arthroplasty within the study period
2. Patients over 20 years old
3. Patients who have received a sufficient explanation, have sufficient understanding, and have given their free written consent.
4. Patients who have passed 2 years or more since their first total hip arthroplasty

Exclusion Criteria:

1. Patients who are judged to be unsuitable as research subjects by the research physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing revision hip arthroplasty within the study period
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of polyethylene wear particles | When tissue sample was collected during THA revision surgery
  counts / g (tissue sample)
Equivalent circle diameter of polyethylene wear particles | When tissue sample was collected during THA revision surgery
  equivalent circle diameter [㎛]
Aspect ratio of polyethylene wear particles | When tissue sample was collected during THA revision surgery
  aspect ratio
Roundness of polyethylene wear particles | When tissue sample was collected during THA revision surgery
  roundness

SECONDARY OUTCOMES:
Body mass index | When tissue sample was collected during THA revision surgery
  kg/m2
Hip joint flexion angle | When tissue sample was collected during THA revision surgery
  Degrees
Hip joint exertion angle | When tissue sample was collected during THA revision surgery
  Degrees
Hip joint adduction angle | When tissue sample was collected during THA revision surgery
  Degrees
Hip joint abduction angle | When tissue sample was collected during THA revision surgery
  Degrees
Hip dysfunction and Osteoarthritis Outcome. Score for Joint Replacement | When tissue sample was collected during THA revision surgery
  0(worse)-100(best)
Harris Hip Score | When tissue sample was collected during THA revision surgery
  0(worse)-100(best)
University of California at Los Angeles activity score | When tissue sample was collected during THA revision surgery
  １(worse)-10(best)

CONTACTS AND LOCATIONS:
Overall Officials: Yukihide Minoda, MD, PhD, Principal Investigator — Osaka Metropolitan University
Locations (2):
- Mayo Clinic, Rochester, Minnesota, United States
- Osaka Metropolitan University, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Iwakiri K, Iwaki H, Kobayashi A, Minoda Y, Kagiyama H, Kadoya Y, Takaoka K. Characteristics of Hylamer polyethylene particles isolated from peri-prosthetic tissues of failed cemented total hip arthroplasties. J Biomed Mater Res B Appl Biomater. 2008 Apr;85(1):125-9. doi: 10.1002/jbm.b.30924. PMID 17806109
- [Result] Hata K, Minoda Y, Ikebuchi M, Mizokawa S, Ohta Y, Miyazaki N, Miyake Y, Nakamura H. In vivo wear particles of remelted highly crosslinked polyethylene after total hip arthroplasty: report of four cases. J Mater Sci Mater Med. 2015 Mar;26(3):133. doi: 10.1007/s10856-015-5472-9. Epub 2015 Feb 25. PMID 25712074
- [Result] Minoda Y, Kobayashi A, Sakawa A, Aihara M, Tada K, Sugama R, Iwakiri K, Ohashi H, Takaoka K. Wear particle analysis of highly crosslinked polyethylene isolated from a failed total hip arthroplasty. J Biomed Mater Res B Appl Biomater. 2008 Aug;86(2):501-5. doi: 10.1002/jbm.b.31048. PMID 18360879